CLINICAL TRIAL: NCT03684525
Title: Assessment of Extraction of Primary Canines in Treating Mesioangular Displaced Permanent Canines Using Cone Beam Computed Tomography (CBCT). A Randomized Controlled Trial
Brief Title: Assessment of Extraction of Primary Canines in Treating Mesioangular Displaced Permanent Canines
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: King Abdulaziz University (Other)
Responsible Party: Principal Investigator, Najlaa Alamoudi, Professor Najlaa Alamoudi, King Abdulaziz University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: KingAbdulazizUniversity
Record Dates: First submitted 2017-10-10; First posted 2018-09-25 (Actual); Last update posted 2018-09-25 (Actual); Status verified 2018-09

CONDITIONS: Displaced Tooth
Keywords: Mesioangular displaced canines; Interceptive treatment

STUDY DESIGN:
Intervention Model Description: Randomized controlled clinical trial following CONSORT guidelines. Patients to be allocated equally to two groups: one treatment group and one control group as follows:
  * Group 1: Extraction of primary maxillary canines group (EG)
  * Group 2: Control group - no extraction (CG)
Who Masked: Investigator
Masking Description: Two investigators unaware of the group to which the patients belong will carry out all the measurements on CBCT scan. One investigator will crop the view of the extraction site to ensure blinding of the other investigator.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Extraction of primary canines only (Experimental): A total of 43 patients with unilateral mesioangular displaced maxillary canines Interceptive treatment: Extraction of both maxillary primary canines will be held at baseline visit At Baseline (T0): Clinical examinatiion + CBCT scan and then both primary canines will be extracted At 6 month follow-up (T1): Clinical examination only At 12 month follow-up: Clinical examination +/- CBCT scan
  Treatment Plan :
  * If displaced canine is not erupted and no improvement in position radiographically is noticed, patient will be referred to orthodontic/oral surgery department
  * If Canine is emerged to oral cavity: No further CBCT scan will be taken
  * If Position of canine is improved radiographically: Follow up untill canine emerges, total observation time is 18 months
  Interventions: Procedure: Extraction of primary canines
- Control group- no extraction (No Intervention): A total of 43 patients with unilateral mesioangular displaced maxillary canines At Baseline (T0): Clinical examinatiion + CBCT scan , no extraction At 6 month follow-up (T1): Clinical examination At 12 month follow-up: Clinical examination +/- CBCT scan
  Treatment Plan :
  * If displaced canine is not erupted and no improvement in position radiographically is noticed, patient will be referred to orthodontic/oral surgery department
  * If Canine is emerged to oral cavity: No further CBCT scan will be taken
  * If Position of canine is improved radiographically: Follow up untill canine emerges, total observation time is 18 months

INTERVENTIONS:
Procedure: Extraction of primary canines — At Baseline (T0): Clinical examinatiion + CBCT scan and then both primary canines will be extracted At 6 month follow-up (T1): Clinical examination only At 12 month follow-up: Clinical examination +/- CBCT scan
  Treatment Plan :
  * If displaced canine is not erupted and no improvement in position radiographically is noticed, patient will be referred to orthodontic/oral surgery department
  * If Canine is emerged to oral cavity: No further CBCT scan will be taken
  * If Position of canine is improved radiographically: Follow up untill canine emerges, total observation time is 18 months
  Arms: Extraction of primary canines only

SUMMARY:
This research project is important because there is no gold standard to rely on regarding the effect of the extraction of primary canines as an interceptive treatment for children with mesioangular displaced canines.

Further investigations are needed to assess the impact of extractions of primary canines approach on the eruption rate or change in position of mesioangular displaced canines by comparing to non-extraction control group in an attempt to overcome the deficiencies in study designs of previously published studies.

DETAILED DESCRIPTION:
Primary objective:

To assess the effect of interceptive extraction of the primary canine on success of eruption of the permanent canine or the change in the position of displaced canine radiographically in children with mesioangular displaced canine when compared to non-extraction control group

Secondary objectives:

1. To evaluate the patient satisfaction and pain experience during treatment
2. To assess the effect of interceptive extraction of the primary canine on the condition of the roots of neighboring teeth
3. To evaluate the effect of stage of root development on the level of correction of permanent canine position radiographically over time when comparing unilateral mesioangular displaced canine subgroup with its contralateral control
4. To identify the effect of independent variables on the outcome of interceptive treatment

Materials and Methods

Study design: Randomized controlled clinical trial following CONSORT guidelines. Patients to be allocated equally to one of the three groups: Two treatment groups and one control group as follows:

* Group 1: Extraction of primary maxillary canine only group (EG)
* Group 2: Control group - no extraction (CG)
* Subgroup of unilateral mesioangular displaced canine vs. contralateral canine as the control group Patients' recruitment will take place in Pediatric Dentistry Speciality Clinic at King Abdulaziz Faculty of Dentistry.

Randomization:

The investigators plan to use a randomized block design, with blocks of varying lengths. The block size will be 6 or 9; the lengths will be randomly chosen, with equal probability, and the length of any given block will be unknown to investigators and clinic personnel. This block design assures balanced allocation into the three groups.

Sample size calculation Based on previously published data (Naoumova et al., 2015); which found 30% difference of displaced canine eruption rates between extraction of canine group (69%) and non-extraction (39%). Based on the alpha significance level of 0.05 and a beta of 0.20 to achieve 80 percent power to detect a 30% differences between groups, two-sided Pearson's chi-square test with normal approximation indicates that 43 patients with unilateral mesioangular displacement were needed in each group for this group comparison.

Given the study design with two groups with equal sample size across groups, hence there will be a total of 43x2=86 patients with unilateral needed in total.

The tooth rather than the patient will be used as the unit of analysis. Inclusion of bilateral mesioangular displaced canines will reduce the number of patients needed; however, one patient with bilateral mesioangular displaced canines cannot be simply counted as two study units in analysis due to high collection within the teeth from the same patient. Adjusting for clustering within patient of bilateral mesioangular displaced canines using the correction by Donner et al. assuming intra patient correlation of 0.5, one bilateral mesioangular displaced canines will be counted as 1.3 study units (2/(1+(2-1)*0.5) (Donner et al., 1981). Naoumova's study had about one third of the patients recruited having bilateral palatally displaced canines, so it is estimated that about 30 patients recruited in this study will have bilateral mesioangular displaced canines, and the contribution of these 30 patients with bilateral mesioangular displaced canines will be equivalent to about 40 patients with unilateral mesioangular displaced canines. These extra (10 study units) contributions from the patients with bilateral mesioangular displaced canines will compensate for possible 10% dropouts during the 12 month study period. Hence, a total of 86 patients (regardless of unilateral or bilateral mesioangular displaced canines will be recruited).

Treatment Process and Intervention:

At baseline (T0), the first CBCT scan will take place and the mesioangular displaced canine position will be precisely localized in three planes. The extraction of the primary canines will be carried out on the same day for the extraction groups.

Six months later the (T1) patients of both groups will undergo a simple clinical examination. At the 12-month follow-up period (T2), a new CBCT scan will be taken if the canine has not yet emerged through the gingival tissue.

Patients with unerupted canines with no improvement in position will be referred to the orthodontic department for combined surgical and orthodontic treatment to be carried out. However, if the position of the canine has improved radiographically, the patient will be clinically followed up until the canine erupts into the oral cavity with a total observation period of 18 months. No further radiographs will be taken.

Alginate impressions for study cast construction will be taken at baseline (T0) prior to extraction, at 6 months (T1), and at 12 months (T2). Space analysis will be performed using Moyers prediction values .

The root development of each mesioangular displaced canine will be assessed by the method developed by Nolla (Nolla, 1960).

Moreover, root development stage of unilateral mesioangular displaced canines subgroup will be measured and compared to normally developing contralateral canine that is considered as its control.

The condition of the roots of neighbouring teeth will be assessed according to the following classification by Ericson and Kurol. Grade 1 no resorption and an intact root surface; Grade 2 slight resorption of up to half of the dentine thickness; Grade 3 is moderate resorption midway to the pulp or more; Grade 4 severe resorption, with the pulp being exposed through the resorption site (Ericson and Kurol, 2000)

Pain experience in extraction groups will be recorded at baseline (T0) after extraction procedure and at 1 week follow up using a questionnaire that will be given to patients about their overall pain experience and discomfort .The questionnaire has been used previously and had acceptable validity and reliability (Feldmann et al., 2007).

Patient satisfaction will also be evaluated at the end of the study by asking the parents to fill patient satisfaction questionnaire. Validation of parent satisfaction questionnaire was done by (Bennett et al., 2001).

Both questionnaires will be translated to Arabic and the validity and reliability will be tested.

Variables

* Independent demographic variables include family history and gender
* Independent clinical variables include presence or absence of crowding, malocclusion classification, presence of peg-shaped/missing laterals, disturbance of eruption sequence , stage of root development and presence of unilateral vs. bilateral mesioangular displaced canine.

Main outcome variables include measurements on CBCT in different views following previously published study which compared the following measurements against measurements on dry skull and concluded that the linear and angular measurements are accurate on CBCT images and are considered valid diagnostic variables (Naoumova et al., 2014).

Measurements will be done using CS 3D imaging Software Carestream Company. The following measurements will be recorded for each CBCT scan:

Linear measurements (mm)

1. Axial view: canine cusp tip- dental arch plane and canine root apex- dental arch plane .

   Dental arch plane is a line that is drawn in the center of the dental arch bisecting teeth present in the arch.
2. Coronal view: Canine cusp tip- midline
3. Sagittal view: The vertical height from canine tip to occlusal line . Occlusal line is a line that will be drawn between the incisal edges of upper and lower incisors.

Angular measurements (°)

1. Frontal (coronal) view: measurement of the mesioangular angle relative to the reference line (fixed line that will be drawn through the hard palate).
2. Sagittal view: measurement of sagittal angle relative to the reference line Blinding Two examiners unaware of the group to which the patients belong will carry out all the measurements on CBCT scan. One examiner will crop the view of the extraction site to ensure blinding of the other examiner.

Reliability on CBCT scan measurements Two independent examiners will carry out all the linear and angular measurements on CBCT scans. Both examiners will undergo CBCT software use training by oral radiologist. Both examiners will undergo a calibration exercise of the measuring technique before starting the trial to ensure inter-examiner reliability. Kappa statistics will be used to calculate inter-examiner reproducibility.

Justification of the use of CBCT in this study

Following the principle of "as low as reasonably achievable" (ALARA); CBCT is justified to be used to detect canine displacement if the field of view (FOV) is small and restricted to the area of interest. The American Academy of Oral and Maxillofacial Radiology supports the safe use of CBCT for diagnosis of anomalies in dental position prior and during treatment if the FOV is small (AAOMR, 2013). When the effective dose (µSv) was measured on a 10-year old phantom, it was found that 6x16 maxillary imaging resulted in significantly lower doses than other fields. The effective dose on the maxilla with FOV 6x16 cm ranged from 4.7-38.7 µSv (Ludlow and Walker, 2013). This wide range of exposure profile depends not only on machine type but also on different technical parameters.

Therefore, investigators are going to do their best effort to minimize the radiation exposure of the patient by controlling every measure in imaging protocols to reduce the radiation dose. This can be achieved by choosing a small field of view 6x16 (cm), by selecting bigger pixels size to get lower resolution,0.4 voxels will be selected for the resolution. QuickScan scanning protocol (seconds) with an acquisition time of 4.8 seconds will be selected . Tube energy (kV) will be 120 KVP and the tube current will be 10 mAs. The total effective dose will be around 22 µSv which is in the range of taking one lateral cephalometric radiograph and one panoramic radiograph combined together (Ludlow et al., 2015).

Statistics

* For primary objectives that assess successful eruption rate: Chi-square or Fisher exact tests will be used to detect differences in rates among groups
* For primary objectives that assess change in position of PDC, one-way ANOVA or t-test will be used (continuous outcome)
* The analyses of secondary objectives will be conducted in the same way. If categorical outcome has more than two levels, logistic regression will be used.
* All data analyses will be conducted with the SAS statistical package.

ELIGIBILITY:
Inclusion Criteria:

The following inclusion (eligibility) criteria have to be fulfilled by the patients participating in the study:

* Age of patients at diagnosis should be between 9 and 12 years old
* Presence of firm maxillary primary canines
* Identification of maxillary unilateral or bilateral mesioangular displaced maxillary canine by clinical examination .
* Canine position will be confirmed by means of horizontal tube shift following Clark's rule using two peripaical radiographs of the canine region.

Exclusion Criteria:

* Any systemic condition, craniofacial syndromes or cleft lip and/or palate.
* Patients with previous or ongoing orthodontic treatment Imaging exclusion criteria will be checked at baseline and follow-up.
* Severe canine displacement according to Power and Short (Power and Short, 1993). This includes complete overlap of the canine relative to adjacent incisor and beyond (Stage 3). Severe angulation relative to the midline. Canine crown vertical height is above the full length of adjacent incisors roots (see index below for illustrations).
* Severe Resorption of adjacent teeth, grade 3 or 4 according to Ericson and Kurol at baseline or during the trial (Ericson and Kurol, 2000).
* Presence of pathology surrounding the canine (such as cyst, supernumerary, odontome).
* Closed apex of mesioangular displaced canine

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 86 (Estimated)
Dates: Start 2017-11-28 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Successful eruption of maxillary permanent canines into the dental arch | 12 months
  The successful outcome is the eruption of maxillary permanent canines within 12 months into the dental arch

SECONDARY OUTCOMES:
Successful improvement of permanent canine position radiographically | 12 months
  At 12 month follow up a new CBCT scan will be taken to check if there will be any improvement in canines position radiographically compared to the CBCT scan that will be taken at baseline

CONTACTS AND LOCATIONS:
Overall Officials: Najlaa M Alamoudi, BDS MSc DSc, Principal Investigator — King Abdulaziz University, Faculty of Dentistry
Locations (1):
- King Abdulaziz University, Dental University Hospital, Jeddah, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] American Academy of Oral and Maxillofacial Radiology. Clinical recommendations regarding use of cone beam computed tomography in orthodontics. [corrected]. Position statement by the American Academy of Oral and Maxillofacial Radiology. Oral Surg Oral Med Oral Pathol Oral Radiol. 2013 Aug;116(2):238-57. doi: 10.1016/j.oooo.2013.06.002. PMID 23849378
- [Background] Bennett ME, Tulloch JF, Vig KW, Phillips CL. Measuring orthodontic treatment satisfaction: questionnaire development and preliminary validation. J Public Health Dent. 2001 Summer;61(3):155-60. doi: 10.1111/j.1752-7325.2001.tb03383.x. PMID 11603319
- [Background] Donner A, Birkett N, Buck C. Randomization by cluster. Sample size requirements and analysis. Am J Epidemiol. 1981 Dec;114(6):906-14. doi: 10.1093/oxfordjournals.aje.a113261. No abstract available. PMID 7315838
- [Background] Ericson S, Kurol J. Incisor root resorptions due to ectopic maxillary canines imaged by computerized tomography: a comparative study in extracted teeth. Angle Orthod. 2000 Aug;70(4):276-83. doi: 10.1043/0003-3219(2000)0702.0.CO;2. PMID 10961776
- [Background] Feldmann I, List T, John MT, Bondemark L. Reliability of a questionnaire assessing experiences of adolescents in orthodontic treatment. Angle Orthod. 2007 Mar;77(2):311-7. doi: 10.2319/0003-3219(2007)077[0311:ROAQAE]2.0.CO;2. PMID 17319767
- [Background] Ludlow JB, Timothy R, Walker C, Hunter R, Benavides E, Samuelson DB, Scheske MJ. Effective dose of dental CBCT-a meta analysis of published data and additional data for nine CBCT units. Dentomaxillofac Radiol. 2015;44(1):20140197. doi: 10.1259/dmfr.20140197. PMID 25224586
- [Background] Ludlow JB, Walker C. Assessment of phantom dosimetry and image quality of i-CAT FLX cone-beam computed tomography. Am J Orthod Dentofacial Orthop. 2013 Dec;144(6):802-17. doi: 10.1016/j.ajodo.2013.07.013. PMID 24286904
- [Background] Naoumova J, Kjellberg H, Palm R. Cone-beam computed tomography for assessment of palatal displaced canine position: a methodological study. Angle Orthod. 2014 May;84(3):459-66. doi: 10.2319/070913-502.1. Epub 2013 Oct 25. PMID 24160995
- [Background] Naoumova J, Kurol J, Kjellberg H. Extraction of the deciduous canine as an interceptive treatment in children with palatal displaced canines - part I: shall we extract the deciduous canine or not? Eur J Orthod. 2015 Apr;37(2):209-18. doi: 10.1093/ejo/cju040. Epub 2014 Sep 22. PMID 25246604
- [Background] NOLLA, C. 1960. The development of the Permanent Teeth. Journal of Dentistry of Children 27, 254-266.